CLINICAL TRIAL: NCT05597007
Title: Virtual Care to Improve Post-Intensive Care Syndrome
Acronym: VPICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hopital Montfort (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20220547-01H
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Post Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Clinic participation
  Interventions: Behavioral: VPICS Clinic

INTERVENTIONS:
Behavioral: VPICS Clinic — Participants will complete a mix of mandatory synchronous and asynchronous sessions with their Health Group to address PICS. Participants will spend 15 minutes daily on physiotherapy, and 15 minutes on cognitive therapy. There are also 2h time slots everyday for participants to join for an optional check-in with their health coach, who can support them in their individual activities. Participants will spend 15 minutes weekly responding to journal prompts about nutrition and general challenges.

SUMMARY:
The goal of this interventional trial is to learn about whether a virtual clinic can help patients with post-intensive care unit syndrome regain functional ability. Participants will participate in a 12-month online clinic where they will receive physiotherapy, nutritional planning, mental health support and cognitive strengthening. Functional capacity will be measured throughout the clinic. After, they will be asked questions about their clinic experience, and complete a questionnaire.

DETAILED DESCRIPTION:
Virtual Care to Improve Post-Intensive Care Syndrome (V-PICS) is a multidisciplinary virtual clinic designed to address the three components of post-intensive care syndrome (PICS): physical impairment, cognitive decline and mental health challenges. This initiative targets ICU survivors who received mechanical ventilation for a minimum of 48 hours. Referred patients will access live sessions with healthcare professionals who will guide at-home strategies to address PICS including physiotherapy, nutritional planning, mental health support and cognitive strengthening. The clinic will provide an integrated approach to addressing the challenges faced by ICU survivors. The feasibility of this virtual clinic will be assessed by measuring patient satisfaction, clinic effectiveness and levels of engagement and attendance. The study's findings will inform the creation of a robust multi-centre clinical trial that will contribute to the creation of a national standard of PICS care and increase health system efficiencies.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* received mechanical ventilation for a minimum of 48 hours in the ICU
* discharged from the hospital in the 2 months prior to study start

Exclusion Criteria:

* Individuals originating from an assisted living/ long-term care facility
* lack a capacity for informed consent
* have end-stage illnesses
* present a significant fall risk
* cannot speak English or French
* do not have the technological skills or caregiver support to ensure digital literacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Creation of a feasible virtual model of PICS care. | Measured at Month 12
  Measured by participant focus groups concerning participation, attrition, adherence, engagement, perceived value.

SECONDARY OUTCOMES:
Participant satisfaction | Measured at Month 12
  Measured by the Canadian Health Care Evaluation Project (CANHELP) survey. The validated questionnaire assesses healthcare satisfaction in elderly patients with life-limiting illnesses. This abbreviated 15-item questionnaire contains questions pertaining to trust in healthcare providers, sense of dignity, quality of communication and confidence in planning for future healthcare needs. Each question has 5 options for level of agreement with a given statement (Not at all, not very, somewhat, very, completely).
Participant satisfaction | Measured at Month 12
  Measured by focus group thematic analysis.
Increased participant quality of life. | Baseline and Month 12
  Measured by the Functional Independence Measure (FIM). The validated FIM consists of 18 questions and addresses six motor and cognitive functional areas. Each element of the FIM is rated on a scale of 1 to 7, with 7 signifying complete independence.
Increased participant quality of life. | Baseline and Month 12
  Measured by the Patient Reported Outcomes Measurement Information System (PROMIS). The PROMIS examines physical function, anxiety, depression, fatigue, sleep disturbance, participation in social roles and activities, pain interference/intensity. The PROMIS-29 questionnaire has 29 questions rated on scales of 1 to 5 or 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Kwadwo Kyeremanteng, MD, Principal Investigator — Hôpital Montfort
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Montfort Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No